CLINICAL TRIAL: NCT04765046
Title: The Influence of Age on EEG Signals and Consciousness During Anesthesia (TIARA)
Brief Title: The Influence of Age on EEG Signals and Consciousness During Anesthesia
Acronym: TIARA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MDT18067TIARA
Record Dates: First submitted 2021-01-08; First posted 2021-02-21 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Anesthesia
Keywords: Bispectral index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BIS™ System (Other): Enrolled subjects who are undergoing a standard of care elective surgery under general anesthesia, will be equipped with the BIS system to non-invasively measure and interpret brain waive activity directly related to the effects of anesthetic agents during the surgery duration.
  Interventions: Device: Bispectral (BIS™) Complete Monitoring System

INTERVENTIONS:
Device: Bispectral (BIS™) Complete Monitoring System — The BIS™ Complete Monitoring System is a user-configurable patient monitoring system designed to monitor the hypnotic state of the brain based on the acquisition and processing of EEG signals. The BIS technology converts raw EEG data acquired from the frontal cortex into a single number to measure the level of consciousness, called the BIS index. A bilateral sensor is to be placed on the patient's forehead to collect the EEG signals and transmit them back to the system.

SUMMARY:
This is a prospective, multi-center, non-invasive, interventional, data collection study to improve the current BIS algorithm in the elderly adult population.

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-invasive, interventional, data collection study to improve the current BIS algorithm in the elderly adult population. The BIS system will be used on-label as approved in the respective study site countries to monitor and non-invasively measure and interpret brain wave activity directly related to the effects of anesthetic agents. The study's purpose is to evaluate the relationship between BIS parameters, age, and depth of anesthesia in patients undergoing surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

A potential subject may be included for participation in the study if the subject has/is:

1. ≥18 years of age
2. American Society of Anesthesiologists (ASA) physical status I-III
3. Able and willing to participate in the study and sign the informed consent form
4. Will undergo non-ambulatory elective surgery under general anesthesia
5. Has an expected surgery time >2 hours

Exclusion Criteria:

A potential subject will be excluded from participating in the study if the subject has/is:

1. Pregnant
2. Unwilling to undergo EEG measurement
3. Undergone brain surgery procedure or had a cerebrovascular accident or severe head trauma in the last 10 years
4. Alcohol or illicit drug use, which prevents normal functioning in society or has led to organ toxicity. Chronic use of opioids, narcotics, or analgesics, which may limit a subject's responsiveness to analgesic dosages.
5. Known or suspected electroencephalograph abnormality (e.g., epilepsy or scarring)
6. Presence of a major psychiatric condition such as Bipolar disorder/ schizophrenia/ Alzheimer's disease/ dementia/ Parkinson's disease /major depression
7. Severe visual or auditory disorder
8. Cannot understand or is unwilling to perform the study assessments, according to the investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Dahan, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (2):
- Rambam Health Care Campus, Haifa, Israel
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kanonidou Z, Karystianou G. Anesthesia for the elderly. Hippokratia. 2007 Oct;11(4):175-7. PMID 19582189
- [Background] Punjasawadwong Y, Phongchiewboon A, Bunchungmongkol N. Bispectral index for improving anaesthetic delivery and postoperative recovery. Cochrane Database Syst Rev. 2014 Jun 17;2014(6):CD003843. doi: 10.1002/14651858.CD003843.pub3. PMID 24937564
- [Background] Glass PS, Bloom M, Kearse L, Rosow C, Sebel P, Manberg P. Bispectral analysis measures sedation and memory effects of propofol, midazolam, isoflurane, and alfentanil in healthy volunteers. Anesthesiology. 1997 Apr;86(4):836-47. doi: 10.1097/00000542-199704000-00014. PMID 9105228
- [Background] Flaishon R, Windsor A, Sigl J, Sebel PS. Recovery of consciousness after thiopental or propofol. Bispectral index and isolated forearm technique. Anesthesiology. 1997 Mar;86(3):613-9. doi: 10.1097/00000542-199703000-00013. PMID 9066327
- [Background] Schwab HS, Seeberger MD, Eger EI 2nd, Kindler CH, Filipovic M. Sevoflurane decreases bispectral index values more than does halothane at equal MAC multiples. Anesth Analg. 2004 Dec;99(6):1723-1727. doi: 10.1213/01.ANE.0000136467.47996.70. PMID 15562061
- [Background] Hans P, Dewandre PY, Brichant JF, Bonhomme V. Comparative effects of ketamine on Bispectral Index and spectral entropy of the electroencephalogram under sevoflurane anaesthesia. Br J Anaesth. 2005 Mar;94(3):336-40. doi: 10.1093/bja/aei047. Epub 2004 Dec 10. PMID 15591328
- [Background] Sengupta S, Ghosh S, Rudra A, Kumar P, Maitra G, Das T. Effect of ketamine on bispectral index during propofol--fentanyl anesthesia: a randomized controlled study. Middle East J Anaesthesiol. 2011 Oct;21(3):391-5. PMID 22428494
- [Background] Alkire MT. Quantitative EEG correlations with brain glucose metabolic rate during anesthesia in volunteers. Anesthesiology. 1998 Aug;89(2):323-33. doi: 10.1097/00000542-199808000-00007. PMID 9710389
- [Background] Werner P, Heinik J, Mendel A, Reicher B, Bleich A. Examining the reliability and validity of the Hebrew version of the Mini Mental State Examination. Aging (Milano). 1999 Oct;11(5):329-34. doi: 10.1007/BF03339808. PMID 10631883
- [Background] Vellas B, Villars H, Abellan G, Soto ME, Rolland Y, Guigoz Y, Morley JE, Chumlea W, Salva A, Rubenstein LZ, Garry P. Overview of the MNA--Its history and challenges. J Nutr Health Aging. 2006 Nov-Dec;10(6):456-63; discussion 463-5. PMID 17183418
- [Background] Perna S, Francis MD, Bologna C, Moncaglieri F, Riva A, Morazzoni P, Allegrini P, Isu A, Vigo B, Guerriero F, Rondanelli M. Performance of Edmonton Frail Scale on frailty assessment: its association with multi-dimensional geriatric conditions assessed with specific screening tools. BMC Geriatr. 2017 Jan 4;17(1):2. doi: 10.1186/s12877-016-0382-3. PMID 28049443
- [Background] Anderson O, Davis R, Hanna GB, Vincent CA. Surgical adverse events: a systematic review. Am J Surg. 2013 Aug;206(2):253-62. doi: 10.1016/j.amjsurg.2012.11.009. Epub 2013 May 1. PMID 23642651

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BIS™ System
Started | 90
Completed | 72
Not Completed | 18
Not completed — Screen Failure | 2
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 4
Not completed — Surgery Cancelled | 8

BASELINE CHARACTERISTICS:
Population: 15 subjects excluded from final analysis due to disqualification of BIS data
Arm/Group | BIS™ System
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (17.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: BIS50
Description: The Bispectral Index (BIS) value, a scale 0-100 with 0 being no brain activity and 100 being fully conscious, at which 50% of subjects are anesthetized at a level they are considered uncounscious based on the MOAA/S score of 0-2
Time Frame: 8 hours
Measure: Mean (95% Confidence Interval); unit: index
Groups:
- Age 18-64: Subjects enrolled aged 18-64
- Age 65+: Subjects enrolled aged 65 and older
Arm/Group | Age 18-64 | Age 65+
Number analyzed (Participants) | 29 | 28
index | 70.9 [67.8 to 73.7] | 74.7 [72.0 to 77.1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment to study exit (directly after completion of data collection during surgery, approximately 8 hours)
Arm/Group | Age 18-64 | Age 65+
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/33
Other Adverse Events (participants affected / at risk) | 0/39 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT04765046/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT04765046/SAP_001.pdf